CLINICAL TRIAL: NCT00752869
Title: Dutasteride in Men Receiving Testosterone Therapy: Impact on Serum PSA, Testosterone, DHT Levels and Prostate Volume: "Implications for Prostate Safety"
Brief Title: Efficacy Study for Use of Dutasteride (Avodart) With Testosterone Replacement
Acronym: DUT/T
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Martin M. Miner, MD, Principal Investigator, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSK 111504; FDA IND # 101,619
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Hypogonadism
Keywords: low testosterone
MeSH Terms: conditions — Hypogonadism | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator): This group will meet the same inclusion and exclusion criteria as the group receiving the study drug
  Interventions: Drug: placebo
- A (Active Comparator): This arm will receive the active medication dutasteride
  Interventions: Drug: dutasteride

INTERVENTIONS:
Drug: dutasteride — 0.5mg by mouth one time per day for 1 year
  Other Names: Avodart; chemical # c27H30F6N202; g1 198745; ind 64,789; code name nda 021319
  Arms: A
Drug: placebo — one tablet per day for 1 year
  Other Names: Inactive substance
  Arms: B

SUMMARY:
This is a study using two FDA approved medications: Testosterone and the study medication, Dutasteride (Avodart 0.5mg/day). Half of the subjects will receive dutasteride and half will receive a placebo. The study medication will be taken for 12 months.

The subjects participating in the study are men who are already taking their own testosterone supplement because they have low testosterone levels which may cause them to experience sexual function difficulties, have fatigue or other symptoms. Testosterone can have an adverse effect of causing an enlarged prostate (Benign Prostatic Hypertrophy) (BPH).

Dutasteride (Avodart) is an approved medication used to decrease the prostate size, prevent urinary symptoms and reduce the risk of surgery.

The researchers would like to see if by taking dutasteride and testosterone at the same time they can prevent the adverse effects of testosterone and at the same time get the positive benefits of testosterone.

There will be 6 scheduled visits for the study and 2 diagnostic tests called a TRUS (TransRectal UltraSound), to evaluate prostate size. The six visits at will include consenting, blood work, two sexual function questionnaires, a physical examination, physical measurements, study medication teaching and dispensing of study medication.

DETAILED DESCRIPTION:
Termination criteria

1. Serum AST or ALT > 3 times ULN
2. Total serum bilirubin > 1.5 times ULN

   * no study termination of a patient with documented Gilberts disease for an isolated bilirubin elevation unless it exceeds 2.5x the upper limit of normal.
3. Hematocrit > 55%
4. Subject experiences any unacceptable or intolerable adverse effect.
5. Subject is non-compliant with the study protocol.
6. Subject needs to take any medication that would interfere with study measurements
7. Subject develops prostate or breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects currently on stable testosterone replacement therapy for 3 months' duration using either the approved transdermal products Androgel® or Testim®, or injections of testosterone enanthate or cypionate with a morning serum testosterone concentration within the normal range (300 - 1000 ng/dl). These will dispensed either by prescription or for injections by the PI or co-PI in the office.
2. Total Serum PSA >1.5 - 10 ng/mL

   * If the total serum PSA is >4ng/mL, the investigator, or a qualified urologist, will perform a 12-core prostate biopsy prior to entry unless such a biopsy has already been performed within the past 6 months.
   * If the PSA rises above 4 during any time of the study, the patient will be referred to urology for biopsy.
   * Patients with any suspicious rise in PSA of >1.0 ng/ml/yr will have a repeat PSA performed within one month of the original value. If the rise in PSA remains >1.0 ng/ml/yr, the patient will undergo a prostate biopsy.
   * b. If the individual has had a negative biopsy more than 6 months previously, with documentation of stable PSA since that time, ie, no sustained increase >1.0ng/ml.
3. Subject is able to read and comprehend the informed consent document.
4. If the subject is on current replacement therapy for hypopituitarism or other multiple endocrine abnormalities, the subject must be on stable doses of thyroid hormone and/or adrenal replacement hormones for at least 14 days prior to enrollment.

Exclusion Criteria:

1. Use of medications including those interactive with dutasteride from prior studies
2. Hematocrit greater than 51%
3. Prostate cancer in men found to have a prostate nodule on initial exam and subsequent positive biopsy
4. No prostate surgery within 2 months of entry
5. No prior use of finasteride, dutasteride within 6 months prior
6. A history of hepatic impairment or abnormal liver function tests (defined as ALT, AST, alkaline phosphatase or bilirubin >1.5 times the upper limit of normal) with the exception that bilirubin elevations up to 2.0 times the upper limit of normal in the presence of normal liver enzymes will be permitted in patients with documented Gilbert's Disease. Subjects with Gilbert's disease not to be excluded.
7. No serum creatinine greater than 2.0 times upper limit of normal
8. No history of alcohol abuse with last 12 months
9. Has received any medication in a clinical trial within 2 months of enrollment
10. Use of anti-androgens, estrogens or coumadin
11. A history or evidence of newly discovered prostate cancer (e.g. positive biopsy or ultrasound, suspicious DRE). In patients with suspicious ultrasound or DRE, including patients with a focal nodule, biopsy shall be performed by a qualified urologist upon study entry unless one was performed and found to be negative within the preceding 6 months.
12. History of or current prostate or breast cancer
13. Baseline EKG with clinically significant abnormal rhythm or abnormal QT interval
14. Systolic blood pressure above 170mmHg or diastolic blood pressure above 90 mm Hg on baseline physical exam
15. Clinically significant peripheral edema on baseline physical exam
16. History of sleep apnea
17. History of psychiatric disorders or major depression
18. Consumption of grapefruit juice within 7 days of enrollment or is unwilling to eliminate use of grapefruit juice during the study period
19. History of allergy to study medication
20. Hemoglobin A1c > 9% in a non-insulin dependent diabetic
21. Subjects with abnormal thyroid function
22. Subjects with significantly elevated triglycerides

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
PSA reduction | with up to 12 months of treatment

SECONDARY OUTCOMES:
PV reduction with up to 12 months of treatment | 1 year treatment
DHT and T levels: serum | 1 year treatment
Prostatic TRUS pre and post treatment | 1 year treatment
IIEF; MHSQ: Questionnaires examining the domains of erectile and orgasmic function in men in the two treatment arms | 1 year treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Miner, MD, Principal Investigator — The Miriam Hospital; Abraham Morgentaler, MD, Principal Investigator — Men's Health Boston
Locations (2):
- United States (2):
  - Men's Health Boston, Boston, Massachusetts
  - The Miriam Hospital, Providence, Rhode Island